CLINICAL TRIAL: NCT05080426
Title: Family Supportive Supervisor Training and Workplace Assessment Tool
Acronym: FSST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Work Life Help (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Ellen Ernst Kossek, Basil S. Turner Distinguished Professor of Management, Work Life Help
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2R42AG050347-02A1 (NIH); 2R42AG050347-02A1 (NIH)
Record Dates: First submitted 2021-08-30; First posted 2021-10-15 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Psychosocial Deprivation; Work-Related Stress; Life-work Imbalance
Keywords: family supportive supervisor behaviors; work-family intervention; supervisor support for family; sick leave; family leave; workplace intervention; work life balance; supervisor training; manager training; work-family conflict; turnover intentions; flexible workplace; psychosocial intervention
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Intervention Model Description: The current study employs a cluster randomization strategy to assign organizations to either Condition A (intervention group) or Condition B (control group). One organization will be randomly assigned to the intervention and the other organization to the control group.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention Group - Managers (Experimental): Mangers in the intervention group will be asked to:
  1. Complete an online survey;
  2. Take the Family Supportive Supervisor Training online (FSST);
  3. Take the Supervisor Support for Leave Use module;
  4. Track their behaviors for two weeks;
  5. Participate in a webinar and have the opportunity to ask questions and give comments;
  6. Complete a post-training survey;
  7. 8-10 managers may also participate in the focus group.
  Interventions: Behavioral: Family Supportive Supervisor Training 2.0
- Control Group - Managers (No Intervention): Managers in the control group will be asked to:
  1. Complete an online survey three times over the course of 5 months.
- Intervention Group - Employees (Experimental): Employees in the intervention group will be asked to:
  1. Complete an online survey three times over the course of 6 months.
  Interventions: Behavioral: Family Supportive Supervisor Training 2.0
- Control Group - Employees (No Intervention): Employees in the control group will be asked to:
  1. Complete an online survey three times over the course of 5 months.

INTERVENTIONS:
Behavioral: Family Supportive Supervisor Training 2.0 — FSST 2.0 is a workplace intervention package designed to increase supervisors' family and leave supportive behaviors and leave supportive behaviors. The package includes Workplace Assessment tool, 2 45-60 minute online training modules (family-supportive supervisor training and supervisors' leave supportive behavior training), a webinar, behavior training, and individualized feedback reports.
  Other Names: FSST 2.0
  Arms: Intervention Group - Employees; Intervention Group - Managers

SUMMARY:
This study will evaluate the effectiveness of FSST 2.0 (family supportive supervisor training plus support for use of family and sick leaves) using a randomized control trial design. We expect the intervention will increase supervisors' family supportive and leave supportive behaviors, which in turn will increase employees' leave use and decrease employees' work-family conflict, emotional exhaustion, depressive symptoms, and turnover intentions. This study will enroll a minimum 200 groups of managers and their employees. Managers in the intervention condition will complete pre- and 2 post-intervention Workplace Assessments, 2 online training modules, 1 webinar where managers can review intervention content and ask questions and share reactions on the materials. Managers in the control group and employees in both groups will complete pre- and 2 post-intervention Workplace Assessments. The post-intervention Workplace Assessment will be completed 3 and 6 months after the intervention. The total duration of the study is 9 months as the wait list control group will be offered the intervention and 2nd follow up survey after the 6-month trial.

DETAILED DESCRIPTION:
This study will evaluate the effectiveness of FSST 2.0 (family supportive supervisor training plus support for use of family and sick leaves) using a randomized control trial design.

* Phase of the Trial Based on the NIH's definition, the current study is a Phase III clinical trial, which usually involves several hundred or more human subjects, for the purpose of evaluating an experimental intervention in comparison with a standard or controlled intervention or comparing two or more existing treatments.
* Type of trial - a randomized-control trial
* Randomization strategy

  * Randomization method The current study employs a cluster randomization strategy to assign organizations to either Condition A (intervention group) or Condition B (control group) for a few key reasons. First, although only the supervisors will receive the training, the effectiveness of the training will be assessed at the employee' level, thereby needing a nested data structure. Second, cluster randomization is effective in reducing contamination (Puffer et al., 2005). Third, when the intervention is offered at a group level, cluster randomization increases the external validity of the results (Donner & Klar, 2000). Within each organization, we will use a balanced group randomization strategy such that there will be an equal number of workgroups/teams/departments in the intervention or control condition. In the event that there is an odd number of such units, a slight imbalance (i.e., groups per condition) will be off by one group, which has minimal impact on statistical power to detect intervention effects.
  * Unit of randomization - organization
  * Allocation ratio - the same number of teams (one supervisor and at least 6 employees) will be recruited in both organization
  * Timing of randomization - before the baseline assessment
  * The statistician of the study will generate and implement the randomization schema.
* Specification of the number of study groups/arms - 2
* Duration of the study intervention - 6 months
* Follow-up period - 3 and 5 months after the intervention
* Name and brief description of study intervention FSST 2.0 is a workplace intervention package designed to increase supervisors' family and leave supportive behaviors and leave supportive behaviors. The package includes Workplace Assessment tool, 2 30-45-minute online training modules (family-supportive supervisor training and supervisors' leave supportive behavior training), a webinar, behavior training, and organizational reports.
* Control group The current trial employs a wait-list control group, "whereby participants will receive the usual care and will later receive the intervention in addition to the usual care" (Kinser & Robins, 2013, p.2).

One or more organization will be randomly assigned to receive the intervention and the other organization(s) will serve as a wait-list control group.

Mangers in the intervention group will be asked to:

1. Complete a baseline online survey.
2. Take the Family Supportive Supervisor Training online (FSST) - http://wlhmodule1.s3-website.us-east-2.amazonaws.com/
3. Take the Supervisor Support for Leave Use module training online - http://wlhmodule2.s3-website.us-east-2.amazonaws.com/
4. Track their behaviors for two weeks
5. Participate in a webinar with the opportunity to ask Q & A and make comments.

7. Complete up to 2 post-training surveys. 8. Focus groups may also be conducted to get feedback on the training after the study is over.

Employees in the control group and employees in both groups will be asked to:

1. Complete a base line and follow up surveys over the course of 5 months.

The wait list control group will be offered the training after the trial is over.

ELIGIBILITY:
Inclusion Criteria:

* To be 18 years and older
* To be a supervisor with at least six employees or an employee of a participating supervisor

Exclusion Criteria:

* There is no exclusion criterion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1175 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen E Kossek, Ph.D., Principal Investigator — Work Life Help LLC
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified data and referenced resources from a publication will be made available by depositing them at dataverse.org. The dataset will include variables used for the publication with an accompanying codebook containing variables labels and codes in XLSX format. Metadata will be prepared as an XML file, which is compliant with the Data Documentation Initiative (DDI) specification.
  The data and metadata from a publication will be made available by the online publication date.
  The location of the public-use data and how to access the data, as well as acknowledgments of the repository and funding source, will be identified in any publications and presentations about these data.
Supporting Information: Analytic Code
Time Frame: The data and metadata from a publication will be made available by the online publication date.
Access Criteria: The data will be deposited and made available through dataverse.org for easy access to qualified researchers and analysts ( i.e., only those affiliated with a university or similar organization that is listed on the Dataverse website as qualified users). The data will be available for use only for research purposes such as replication and secondary studies. User registration will be required in order to access or download files from dataverse.org.
URL: http://dataverse.org

REFERENCES:
- [Background] Barnett, R. C., Brennan, R. T., & Gareis, K. C.. A closer look at the measurement of Burnout. Journal of Applied Biobehavioral Research.1999; 4(2), 65-78.
- [Background] Boroff, K E, & Lewin, D Loyalty, voice, and intent to exit a union firm: A conceptual and empirical analysis. Industrial and Labor Relations Review. 1997; 51(1), 50-63.
- [Background] Cammann, C., Fichman, M., Jenkins, G. D., & Klesh, J. Michigan Organizational Assessment Questionnaire.1983. In S. E. Seashore, E. E. Lawler, P. H. Mirvis, & C. Cammann (Eds.), Assessing organizational change: A guide to methods, measures, and practices, (pp. 71-138). New York: Wiley-Interscience
- [Background] Carlson, DS, Kacmar, KM, Wayne, JH, & Grzwacz, JG Measuring the positive side of the work-family interface: Development and validation of a work-family enrichment scale. Journal of Vocational Behavior. 2006. 68, 131-164. doi:10.1016/j.jvb.2005.02.002
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Griffin, MA, Neal, A, & Parker, SK. A new model of work role performance: Positive behavior in uncertain and interdependent contexts. 2007; Academy of Management Journal, 50(2), 327-347.
- [Background] Hammer LB, Ernst Kossek E, Bodner T, Crain T. Measurement development and validation of the Family Supportive Supervisor Behavior Short-Form (FSSB-SF). J Occup Health Psychol. 2013 Jul;18(3):285-96. doi: 10.1037/a0032612. Epub 2013 Jun 3. PMID 23730803
- [Background] Hobfoll, SE, Vinokur, AD, Pierce, PF, & Lewandowski-Romps, L. The combined stress of family life, work, and war in Air Force men and women: A test of conservation of resources theory. International Journal of Stress Management. 2012; 19(3), 217-237.
- [Background] Kessler RC, Barker PR, Colpe LJ, Epstein JF, Gfroerer JC, Hiripi E, Howes MJ, Normand SL, Manderscheid RW, Walters EE, Zaslavsky AM. Screening for serious mental illness in the general population. Arch Gen Psychiatry. 2003 Feb;60(2):184-9. doi: 10.1001/archpsyc.60.2.184. PMID 12578436
- [Background] Kossek, EE, Ruderman, MN, Braddy, PW, & Hannum, KM Work-nonwork boundary management profiles: A person-centered approach. Journal of Vocational Behavior.2012; 81, 112-128. doi:10.1016/j.jvb.2012.04.003
- [Background] Kossek, EE, Colquitt, JA, & Noe, RA. Caregiving decisions, well-being, and performance: The effects of place and provider as a function of dependent type and work-family climates, Academy of Management Journal.2001; 44(1), 29-44.
- [Background] Matthews RA, Kath LM, Barnes-Farrell JL. A short, valid, predictive measure of work-family conflict: item selection and scale validation. J Occup Health Psychol. 2010 Jan;15(1):75-90. doi: 10.1037/a0017443. PMID 20063960
- [Background] Matthews, RA, Pineault, L, & Hong, YH. Normalizing the use of single-item measures. Validation of the single-item compendium for organizational psychology, Journal of Business and Psychology. 2022; Doi:10.1007/s10869-022-09813-3
- [Background] Thomas, LT, & Ganster, DC. Impact of family-supportive work variables on work-family conflict and strain: A control perspective. Journal of Applied Psychology. 1995; 80(1), 6-15.
- [Background] Yoon, J, , Lim, J. Organizational support in the workplace: The case of Korean hospital employees. Human Relations. 1999; 82, 923-945.
- [Background] Kossek, E. E., Lawson, K. M., Hammer, L. B., Allen, S., Bodner, T., Perry, M., & Xu, J. (April, 2024). Supervisor support for family/sick leaves intervention: An organizational field experiment. Paper presented at the Society for Industrial and Organizational Psychology (SIOP), Conference, Chicago, IL.
- [Background] Kossek, E. E., Lawson, K. M., Hammer, L. B., Bodner, T., Perry, M., Xu, J., & Allen, S. (June, 2024). Leaders and leaves: Validating and evaluating a new measure of paid family supportive supervisor behaviors for family and sick leave. In E. E. Kossek (Chair), Fostering family supportive work scheduling (or not): Links to family and work outcomes. Symposium presented at the Work Family Researchers Network Conference, Montreal, Canada.

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Organization
Groups:
- Intervention Group - Managers and Employees: Mangers in the intervention group will be asked to:
  1. Complete an online survey;
  2. Take the Family Supportive Supervisor Training online (FSST);
  3. Take the Supervisor Support for Leave Use module;
  4. Track their behaviors for two weeks;
  5. Participate in a webinar and have the opportunity to ask questions and give comments;
  6. Complete a post-training survey;
  7. 8-10 managers may also participate in the focus group.
  Employees in the intervention group were asked to:
  1. Complete an online survey three times over the course of 5 months.
  Family Supportive Supervisor Training 2.0: FSST 2.0 is a workplace intervention package designed to increase supervisors' family and leave supportive behaviors and leave supportive behaviors. The package includes Workplace Assessment tool, 2 45-60 minute online training modules (family-supportive supervisor training and supervisors' leave supportive behavior training), a webinar, behavior training, and individualized feedback reports.
- Control Group - Managers and Employees: Managers in the control group will be asked to:
  1. Complete an online survey three times over the course of 5 months.
  Employees in the control group will be asked to:
  1. Complete an online survey three times over the course of 5 months.
Period: Overall Study
Arm/Group | Intervention Group - Managers and Employees | Control Group - Managers and Employees
Started | 802; 1 Organization | 132; 1 Organization
Managers | 172; 1 Organization | 80; 1 Organization
Employees | 630; 1 Organization | 52; 1 Organization
Completed (Completed at least 1 survey in the study.) | 802; 1 Organization | 132; 1 Organization
Not Completed | 0; 0 Organization | 0; 0 Organization

BASELINE CHARACTERISTICS:
Population: Participants were invited to complete follow-up surveys, even if they did not complete the baseline surveys. The sample size reported in the "Participant Flow" section includes all managers and employees who completed at least 1 of the 3 surveys. The baseline analysis information only includes participants who completed the baseline survey (which is a smaller sample than those included in the "Participant Flow" section).
Groups:
- Intervention Group - Employees: Employees in the intervention group will be asked to:
  1. Complete an online survey three times over the course of 5 months.
  Family Supportive Supervisor Training 2.0: FSST 2.0 is a workplace intervention package designed to increase supervisors' family and leave supportive behaviors and leave supportive behaviors. The package includes Workplace Assessment tool, 2 45-60 minute online training modules (family-supportive supervisor training and supervisors' leave supportive behavior training), a webinar, behavior training, and individualized feedback reports.
- Total: Total of all reporting groups
Arm/Group | Intervention Group - Managers | Control Group - Managers | Intervention Group - Employees | Control Group - Employees | Total
Number analyzed (Participants) | 134 | 52 | 492 | 202 | 880
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.74 (8.74) | 50.78 (7.80) | 44.91 (11.06) | 49.04 (11.17) | 46.93 (10.84)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Men | 31 | 21 | 114 | 56 | 222
  Women | 101 | 31 | 367 | 144 | 643
  Gender Nonconforming | 0 | 0 | 1 | 0 | 1
  Not Reported | 2 | 0 | 10 | 2 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 0 | 112 | 8 | 138
  Not Hispanic or Latino | 116 | 52 | 376 | 194 | 738
  Unknown or Not Reported | 0 | 0 | 4 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 0 | 2
  Asian | 17 | 2 | 86 | 8 | 113
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 3 | 0 | 3
  Black or African American | 30 | 4 | 100 | 17 | 151
  White | 64 | 45 | 184 | 156 | 449
  More than one race | 5 | 0 | 36 | 8 | 49
  Unknown or Not Reported | 17 | 1 | 82 | 13 | 113
Region of Enrollment [Number; unit: participants]
  United States | 134 | 52 | 492 | 202 | 880

OUTCOME MEASURES:

1. Primary Outcome: Change in Family Supportive Supervisor Behaviors
Description: Family supportive supervisor behavior scale. Original scale: Minimum value = 1, Maximum value = 5. Reported numbers represent change in these values over time: Time 3 (5-months post-baseline survey) - Time 1 (baseline survey) scores.
  Positive scores = increase in scores over time (better outcome). Negative scores = decrease in scores over time (worse outcome).
Time Frame: 5 months after the intervention
Population: Employees of trained managers who completed at least one out of three surveys (baseline, 3-month follow-up, 5-month follow-up). Employees could complete follow-up surveys, even if they did not complete the baseline survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group - Employees | Control Group - Employees
Number analyzed (Participants) | 630 | 293
units on a scale | -.08 (.78) | .06 (.79)

2. Primary Outcome: Change in Leave Supportive Supervisor Behaviors
Description: Original scale: Minimum value = 1, Maximum value = 5. Reported numbers represent change in these values over time: Time 3 (5-months post-baseline survey) - Time 1 (baseline survey) scores.
  Positive scores = increase in scores over time (better outcome). Negative scores = decrease in scores over time (worse outcome).
Time Frame: 5 months after the intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intervention Group - Employees: Employees in the intervention group will be asked to:
  1. Complete an online survey three times over the course of 6 months.
  Family Supportive Supervisor Training 2.0: FSST 2.0 is a workplace intervention package designed to increase supervisors' family and leave supportive behaviors and leave supportive behaviors. The package includes Workplace Assessment tool, 2 45-60 minute online training modules (family-supportive supervisor training and supervisors' leave supportive behavior training), a webinar, behavior training, and individualized feedback reports.
Arm/Group | Intervention Group - Employees | Control Group - Employees
Number analyzed (Participants) | 630 | 293
units on a scale | .04 (.65) | -.07 (.53)

3. Secondary Outcome: Change in Work-family Conflict
Description: Work family conflict scale. Original scale: Minimum value = 1, Maximum value = 5. Reported numbers represent change in these values over time: Time 3 (5-months post-baseline survey) - Time 1 (baseline survey) scores.
  Positive scores = increase in scores over time (worse outcome). Negative scores = decrease in scores over time (better outcome).
Time Frame: 5 months after the intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Control Group - Employees: Managers and employees in the control group will be asked to:
  1. Complete an online survey three times over the course of 6 months.
Arm/Group | Intervention Group - Employees | Control Group - Employees
Number analyzed (Participants) | 630 | 293
units on a scale | .03 (.81) | -.04 (.70)

4. Secondary Outcome: Change in Emotional Exhaustion
Description: Emotional exhaustion scale. Original scale: Minimum value = 1, Maximum value = 5. Reported numbers represent change in these values over time: Time 3 (5-months post-baseline survey) - Time 1 (baseline survey) scores.
  Positive scores = increase in scores over time (worse outcome). Negative scores = decrease in scores over time (better outcome).
Time Frame: 5 months after the intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group - Employees | Control Group - Employees
Number analyzed (Participants) | 630 | 293
units on a scale | -.01 (1.33) | -.38 (1.17)

5. Secondary Outcome: Change in Employee's Leave Use
Description: Number of days of leave used for sick or family leave in the past 6 months. Reported numbers represent change in these values over time: Time 3 (5-months post-baseline survey) - Time 1 (baseline survey) scores.
  Positive scores = increase in scores over time. Negative scores = decrease in scores over time.
  Note: higher scores do not represent better or worse outcomes. They are descriptions of use needed for sick or family leave.
Time Frame: 5 months after the intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention Group - Employees | Control Group - Employees
Number analyzed (Participants) | 630 | 293
days | .69 (18.32) | -.32 (11.28)

6. Secondary Outcome: Change in Turnover Intentions
Description: Turnover intentions scale. Original scale: Minimum value = 1, Maximum value = 5. Reported numbers represent change in these values over time: Time 3 (5-months post-baseline survey) - Time 1 (baseline survey) scores.
  Positive scores = increase in scores over time (worse outcome). Negative scores = decrease in scores over time (better outcome).
Time Frame: 5 months after the intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group - Employees | Control Group - Employees
Number analyzed (Participants) | 630 | 293
units on a scale | .03 (.83) | -.06 (.90)

7. Secondary Outcome: Change in Control Over Work
Description: Control over work scale. Original scale: Minimum value = 1, Maximum value = 5. Reported numbers represent change in these values over time: Time 3 (5-months post-baseline survey) - Time 1 (baseline survey) scores.
  Positive scores = increase in scores over time (better outcome). Negative scores = decrease in scores over time (worse outcome).
Time Frame: 5 months after the intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group - Employees | Control Group - Employees
Number analyzed (Participants) | 630 | 293
units on a scale | -.07 (.72) | -.08 (.59)

8. Secondary Outcome: Change in Boundary Countrol
Description: Boundary control scale. Original scale: Minimum value = 1, Maximum value = 5. Reported numbers represent change in these values over time: Time 3 (5-months post-baseline survey) - Time 1 (baseline survey) scores.
  Positive scores = increase in scores over time (better outcome). Negative scores = decrease in scores over time (worse outcome).
Time Frame: 5 months after the intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group - Employees | Control Group - Employees
Number analyzed (Participants) | 630 | 293
units on a scale | .02 (.87) | -.09 (.76)

9. Secondary Outcome: Change in Work-life Climate
Description: Work-life climate scale. Original scale: Minimum value = 1, Maximum value = 5. Higher scores = expected to make more family sacrifices. Reported numbers represent change in these values over time: Time 3 (5-months post-baseline survey) - Time 1 (baseline survey) scores.
  Positive scores = increase in scores over time (worse outcome). Negative scores = decrease in scores over time (better outcome).
Time Frame: 5 months after the intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group - Employees | Control Group - Employees
Number analyzed (Participants) | 630 | 293
units on a scale | .04 (.91) | -.12 (.95)

10. Secondary Outcome: Change in Work-to-family Positive Spillover
Description: WTF positive spillover scale. Original scale: Minimum value = 1, Maximum value = 5. Reported numbers represent change in these values over time: Time 3 (5-months post-baseline survey) - Time 1 (baseline survey) scores.
  Positive scores = increase in scores over time (better outcome). Negative scores = decrease in scores over time (worse outcome).
Time Frame: 5 months after the intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group - Employees | Control Group - Employees
Number analyzed (Participants) | 630 | 293
units on a scale | .05 (.71) | .06 (.68)

11. Secondary Outcome: Change in General Supervisor Support
Description: General supervisor support scale. Original scale: Minimum value = 1, Maximum value = 5. Reported numbers represent change in these values over time: Time 3 (5-months post-baseline survey) - Time 1 (baseline survey) scores.
  Positive scores = increase in scores over time (better outcome). Negative scores = decrease in scores over time (worse outcome).
Time Frame: 5 months after the intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group - Employees | Control Group - Employees
Number analyzed (Participants) | 630 | 293
units on a scale | -.10 (.70) | -.08 (.69)

12. Secondary Outcome: Change in Supervisor Performance Support
Description: Supervisor performance support scale. Original scale: Minimum value = 1, Maximum value = 5. Reported numbers represent change in these values over time: Time 3 (5-months post-baseline survey) - Time 1 (baseline survey) scores.
  Positive scores = increase in scores over time (better outcome). Negative scores = decrease in scores over time (worse outcome).
Time Frame: 5 months after the intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group - Employees | Control Group - Employees
Number analyzed (Participants) | 630 | 293
units on a scale | .02 (.75) | -.02 (.85)

13. Secondary Outcome: Change in Job Satisfaction
Description: Job satisfaction scale. Original scale: Minimum value = 1, Maximum value = 5. Reported numbers represent change in these values over time: Time 3 (5-months post-baseline survey) - Time 1 (baseline survey) scores.
  Positive scores = increase in scores over time (better outcome). Negative scores = decrease in scores over time (worse outcome).
Time Frame: 5 months after the intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group - Employees | Control Group - Employees
Number analyzed (Participants) | 630 | 293
units on a scale | -.03 (.68) | -.04 (.54)

14. Secondary Outcome: Change in Job Performance
Description: Job performance scale. Original scale: Minimum value = 1, Maximum value = 5. Reported numbers represent change in these values over time: Time 3 (5-months post-baseline survey) - Time 1 (baseline survey) scores.
  Positive scores = increase in scores over time (better outcome). Negative scores = decrease in scores over time (worse outcome).
Time Frame: 5 months after the intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group - Employees | Control Group - Employees
Number analyzed (Participants) | 630 | 293
units on a scale | -.05 (.52) | .07 (.43)

15. Secondary Outcome: Change in Organizational Commitment
Description: Organizational commitment item. Original scale: Minimum value = 1, Maximum value = 5. Reported numbers represent change in these values over time: Time 3 (5-months post-baseline survey) - Time 1 (baseline survey) scores.
  Positive scores = increase in scores over time (better outcome). Negative scores = decrease in scores over time (worse outcome).
Time Frame: 5 months after the intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group - Employees | Control Group - Employees
Number analyzed (Participants) | 630 | 293
units on a scale | -.03 (.87) | -.03 (.82)

16. Secondary Outcome: Change in Perceived Health
Description: Perceived health item. Original scale: Minimum value = 1, Maximum value = 5. Higher scores = better health. Reported numbers represent change in these values over time: Time 3 (5-months post-baseline survey) - Time 1 (baseline survey) scores.
  Positive scores = increase in scores over time (better outcome). Negative scores = decrease in scores over time (worse outcome).
Time Frame: 5 months after the intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group - Employees | Control Group - Employees
Number analyzed (Participants) | 630 | 293
units on a scale | .02 (.47) | .01 (.47)

17. Secondary Outcome: Change in Psychological Distress
Description: Psychological distress scale. Original scale: Minimum value = 1, Maximum value = 5. Reported numbers represent change in these values over time: Time 3 (5-months post-baseline survey) - Time 1 (baseline survey) scores.
  Positive scores = increase in scores over time (worse outcome). Negative scores = decrease in scores over time (better outcome).
Time Frame: 5 months after the intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group - Employees | Control Group - Employees
Number analyzed (Participants) | 630 | 293
units on a scale | -.09 (.64) | -.10 (.43)

18. Secondary Outcome: Change in Perceived Stress
Description: Perceived stress scale. Original scale: Minimum value = 1, Maximum value = 5. Reported numbers represent change in these values over time: Time 3 (5-months post-baseline survey) - Time 1 (baseline survey) scores.
  Positive scores = increase in scores over time (worse outcome). Negative scores = decrease in scores over time (better outcome).
Time Frame: 5 months after the intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group - Employees | Control Group - Employees
Number analyzed (Participants) | 630 | 293
units on a scale | .02 (.66) | -.03 (.52)

ADVERSE EVENTS:
Time Frame: 5 months
Description: Supervisors undergoing the training could experience stress from recalling or experiencing challenging interactions that could occur between supervisors and employees regarding managing of the leave or their own family or personal need for sick leave and their supervisors support. Employees completing the survey on supervisor support could recall stress related to disclosure of the need for leaves or less supportive supervisor interactions for requesting policy use.
Arm/Group | Intervention Group - Managers | Control Group - Managers | Intervention Group - Employees | Control Group - Employees
All-Cause Mortality (participants affected / at risk) | 0/172 | 0/80 | 0/630 | 0/293
Serious Adverse Events (participants affected / at risk) | 0/172 | 0/80 | 0/630 | 0/293
Other Adverse Events (participants affected / at risk) | 0/172 | 0/80 | 0/630 | 0/293

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-10): https://cdn.clinicaltrials.gov/large-docs/26/NCT05080426/Prot_SAP_000.pdf